CLINICAL TRIAL: NCT05969808
Title: Effects of Adapted Physical Activities on Visual Motor Integration in Children With Developmental Delay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/ RCR & AHS/23/0726
Record Dates: First submitted 2023-07-23; First posted 2023-08-01 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Development Delay
Keywords: Visual motor integration
MeSH Terms: conditions — Learning Disabilities | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized control trial will be conducted with sample size 30, used to compare the effectiveness of adaptive physical activity on visual motor integration in children with developmental delay. subjects with developmental delay meeting the predetermined inclusion and exclusion criteria will be divided into two groups using non-probability convenient sampling. pre and post assessment will be done by Box and Block Test, Box and Ball Test, Discrete horizontal finger tapping test, Discrete vertical finger tapping with ball and continuous Vertical tapping with ball. subjects in group A will receive Baseline therapy and conventional therapy and group B will receive baseline therapy and adaptive physical activity.
Who Masked: Participant
Masking Description: participants will get separate treatment protocols and possible efforts will be put to mask the both groups about their treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): The control group will participate in regular activities and routines typically provided to children with developmental delays. These activities may include general playtime, basic gross motor activities, and free play with toys for 3 times a week for 45mins for 12 weeks. The control group will not receive any specific intervention targeted at improving visual motor integration, manual dexterity, or intra-limb coordination.
  Experimental group
  Interventions: Other: baseline therapy and conventional therapy
- experimental group (Active Comparator): The Experimental group will receive the baseline treatment as Control group. Adaptive Physical Activities will perform for to improve Visual Motor Integration 3 times a week for 45mins for 12 weeks. Pre and post assessment will be performed by using box and boll test, box and block test, Discrete Vertical Finger Tapping Test (DVFTT), discrete horizontal finger tapping test and discrete vertical tapping test with ball.
  Interventions: Other: baseline treatment and adaptive physical activity

INTERVENTIONS:
Other: baseline therapy and conventional therapy — These activities included were warm-up activities, general playtime, basic gross motor activities, and free play with toys three times a week for 45 minutes for a period of 12 weeks.
  Other Names: control group
  Arms: control group
Other: baseline treatment and adaptive physical activity — The experimental group's intervention plan had the following 12 elements . Each of which was completed for 10 minutes with two-minute breaks. Warm-up activities, puzzles and manipulatives, e.g., interlocking blocks or shape sorting toys, Balloon Badminton, Obstacle course (crawl in Tunnel ), Peg board play, Tactile sensory bin exploration filled with sand, Ball roll and catch, Tracing shapes, Play dough and clay activities, Cutting and pasting.
  Other Names: experimental group
  Arms: experimental group

SUMMARY:
Developmental delay occurs when a child does not achieve developmental milestones in comparison to peers of the same age range. Children and adolescents with developmental delay often experience participation restrictions. Visual motor integration (VMI) is the ability of the child's hands and eyes to work together to guide their movements. Visual motor integration is a broad term encompasses cognitive as well as manual domains. This study will focused on the Manual Dexterity and intra-limb coordination (VMI). And it will evaluate the effects of adaptive physical activity on Visual Motor Integration.

Adaptive physical activities (APAs) are exercises and games that have been specially designed to fulfil the unique needs and skills of special needs or developmental delays.

DETAILED DESCRIPTION:
Randomized control trial will be conducted with sample size 30, used to compare the effectiveness of adaptive physical activity on visual motor integration in children with developmental delay. subjects with developmental delay meeting the predetermined inclusion and exclusion criteria will be divided into two groups using non-probability convenient sampling. pre and post assessment will be done by Box and Block Test, Box and Ball Test, Discrete horizontal finger tapping test, Discrete vertical finger tapping with ball and continuous Vertical tapping with ball. subjects in group A will receive Baseline therapy and conventional therapy and group B will receive baseline therapy and adaptive physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Age group 3-6 (both Gender Male & Female) (39)
* Gross Motor Function Classification System, Level I
* & II (45)
* Manual Ability Classification System (MACS) levels
* 1-3 (46)
* Pre assessed Developmental delayed.

Exclusion Criteria:

* Visually impaired Child
* Children with co-morbidities such as Epilepsy, Hydrocephalus
* Fractures, contractures or conflicting concurrent treatment impacting motor Functioning
* Children with significant cognitive impairments.
* Children who have received specific interventions targeting Visual motor integration, manual dexterity or intra-limb coordination

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
Box and Block Test (BBT) | 12 weeks
  A frequently used assessment test, the Box and Block Test, measure manual dexterity and functional ability, mainly in those with upper limb disabilities. This test measures the capacity to handle items and carry out tasks that call for fine motor abilities(47). 150 tiny wood cubic blocks (1-inch) plus a box with two compartments separated by a wooden wall make up the BBT. 2.5 cm wooden block on each side and a wooden box (53.7 x 25.4 cm) separated into two compartments by a wall 15.2 cm high were the materials used to evaluate the BB test. The BBT entails moving as many little blocks as possible, one at a time, from the compartment on the tested side to the other with the same hand, being careful to cross over the gap. The number of blocks that are correctly shifted in 60 seconds is used to calculate the score
Box and ball test ( BBT) | 12 weeks
  The BBLT followed the same procedure as the BBTs. The sole modification was that the BBLT evaluated the quantity of boccia balls rather than blocks. Due to the size of the compartments, only six balls could fit inside at once. It will be necessary to have two researchers, one at each end of the table.
discrete horizontal finger tapping test (DHFTT) | 12 weeks
  This test used to measure the intra-limb coordination of upper limb.Participants will sit on their chairs and will be placed parallel to a table, at 10 cm from the edge of the tapping plates. The table will be adjusted so that the bottom of the table will be aligned with the players' hips (greater trochanter), and the shoulders of the players' throwing arms with the plate A (start position). Participants will asked to place their non-throwing arm across their chest and keep their throwing hand closed with the index finger extended To complete the test, participants will need to complete 10 tapping cycles, reporting their performance as the average score of the 10 tapping cycles. A cycle was composed of the participants releasing from plate A to hit the plate B (finish position) as fast as possible. The plates were displaced horizontally, and the distance between both plates' centers was 30 cm. The metal plates were 30 cm long by 20 cm wide.
Discrete vertical tapping test with ball | 12 weeks
  this test used to measure the intra-limb coordination. The plates will be arranged vertically in an "L" shape (90°), where plate A will be kept on horizontal but plate B will be placed on the vertical edge .The distance between both plates' centers will be 30 cm, like in the DHFTT, and the two tests will use the same protocol.
continuous vertical tapping test with ball | 12 weeks
  this test used to measure the intra-limb coordination of upper limb. Participants will perform a continuous movement consisting of grasping the ball and hitting plates A and B alternatively as fast as possible within 1 min. Ball contact could be made on any part of the plates.

CONTACTS AND LOCATIONS:
Overall Officials: Laraib Batool, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zapata-Figueroa V, Ortiz-Corredor F. Assessment of Manual Abilities Using the Box and Block Test in Children with Bilateral Cerebral Palsy. Occup Ther Int. 2022 Feb 22;2022:9980523. doi: 10.1155/2022/9980523. eCollection 2022. PMID 35281716